CLINICAL TRIAL: NCT04105738
Title: Voice Analysis as a Predictor for Difficult Intubations
Status: Terminated | Type: Observational
Why Stopped: Terminated: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention.
Sponsor: J. Matthias Walz (Other)
Responsible Party: Sponsor-Investigator, J. Matthias Walz, Principal Investigator, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Other Study IDs: H00012814
Record Dates: First submitted 2019-08-24; First posted 2019-09-26 (Actual); Results first posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia; Difficult Intubation; Difficult Airway Intubation; Speech Dysfunction; Surgery
Keywords: Difficult Intubation; Preoperative Surgical Assessment; Speech Dysfunction; Difficult Airway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Difficult airways: Documented history of difficult airways.
- Control (Not difficult airways): Age matched with normal airways to be used as controls

SUMMARY:
To investigate if signal processing can detect subtle changes in speech production clinically relevant to oropharynx anatomy that may provide an objective measure in the assessment of the presumed difficulty of intubation.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether changes in phonation (sounds coming from vocal cords that occur when a person speaks) can be used as a reliable measure to predict airways that may be difficult to manage in the operating room.

One of the reasons the Preoperative Surgical Assessment (PSE) is performed is to assess subjects for signs of a difficult airway. At this time, none of the assessments have proven to be both highly sensitive and specific. Multiple studies have shown that specific characteristics of a subject's speech can suggest that they may have an issue with the anatomy of the oropharynx (the area consisting of the back of the throat to the vocal cords). Prior research has shown that studying velar vowel sounds, those vowels that require the use of the back of the tongue to pronounce, can be used to predict a disorder called obstructive sleep apnea (a disease associated with difficulty breathing).

The Investigators are trying to determine whether the development of a simple voice study conducted during the PSE visit could alert the Anesthesiologist caring for the subject in the operating room to use the extra precautions provided for people who have a documented history of a difficult airway. It is hoped that the voice analysis test being developed in this study will have the ability to objectively predict a difficult airway for future patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to provide informed consent
* A known documented history of having a difficult airway
* An age-matched control subject with normal airways.

Exclusion Criteria:

* Unable to consent for themselves
* Non-English speaking subjects
* Pregnant Subjects
* Previous Vocal Cord Surgery
* Previous Head and neck surgery that would alter anatomy of hypopharynx

We will not include:

* Prisoners
* Pregnant women
* Individuals who are not yet adults (infants, children, teenagers)
* Adults unable to consent
* Adults who cannot speak English We will not be enrolling subjects who cannot speak English. The subjects must be able to understand the research team member who is testing them as well as the research paradigm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with a documented history of difficult airways and subjects of the same age (matched for age) with normal airways to be used as controls. Patient are labeled as a difficult airway during their hospitalization, they are given a copy of the difficult airway documentation so the patient should be aware already that they are labeled as a difficult airway.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. M Walz, MD, Principal Investigator — UMASS Medical School
Locations (1):
- UMASS Memorial - Medical School Campus, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Asai T, Koga K, Vaughan RS. Respiratory complications associated with tracheal intubation and extubation. Br J Anaesth. 1998 Jun;80(6):767-75. doi: 10.1093/bja/80.6.767. PMID 9771306
- [Background] Moller JT, Johannessen NW, Espersen K, Ravlo O, Pedersen BD, Jensen PF, Rasmussen NH, Rasmussen LS, Pedersen T, Cooper JB, et al. Randomized evaluation of pulse oximetry in 20,802 patients: II. Perioperative events and postoperative complications. Anesthesiology. 1993 Mar;78(3):445-53. doi: 10.1097/00000542-199303000-00007. PMID 8457045
- [Background] Rose DK, Cohen MM. The airway: problems and predictions in 18,500 patients. Can J Anaesth. 1994 May;41(5 Pt 1):372-83. doi: 10.1007/BF03009858. PMID 8055603
- [Background] Fiz JA, Morera J, Abad J, Belsunces A, Haro M, Fiz JI, Jane R, Caminal P, Rodenstein D. Acoustic analysis of vowel emission in obstructive sleep apnea. Chest. 1993 Oct;104(4):1093-6. doi: 10.1378/chest.104.4.1093. PMID 8404173
- [Background] Robb MP, Yates J, Morgan EJ. Vocal tract resonance characteristics of adults with obstructive sleep apnea. Acta Otolaryngol. 1997 Sep;117(5):760-3. doi: 10.3109/00016489709113474. PMID 9349877

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Difficult Airways | Control (Not Difficult Airways)
Started | 13 | 0
Completed | 13 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Terminated: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Difficult Airways | Control (Not Difficult Airways) | Total
Number analyzed (Participants) | 13 | 0 | 13
Age, Continuous [Mean (Full Range); unit: years] | 59 [48 to 72] |  | 59 [48 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 8 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 13 | 0 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 |  | 13

OUTCOME MEASURES:

1. Primary Outcome: Audio Samples to Predict Difficult Intubation
Description: An audio sample from each participant will be broken down into its signal components using signal-processing methods to evaluate whether there are differences between the two participant groups which may correlate to difficult intubation.
Time Frame: 15-20 minutes
Population: Terminated: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention. Signal processing of the audio samples did not work as anticipated and could not be abstracted or analyzed. Additionally, not enough participants were enrolled, including lack of enrollment to the control group, to analyze data.
Arm/Group | Difficult Airways | Control (Not Difficult Airways)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during study participation of 1 day.
Description: Below minimal risk study and participation of 1 day resulted in no adverse events.
Arm/Group | Difficult Airways | Control (Not Difficult Airways)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/0
Other Adverse Events (participants affected / at risk) | 0/13 | 0/0

LIMITATIONS AND CAVEATS:
Due to technical issues, audio recording could not be uploaded or analyzed as anticipated/planned for study, and enrollment did not meet expectations. Therefore, no analysis or results for the study are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/38/NCT04105738/Prot_SAP_000.pdf